CLINICAL TRIAL: NCT03375424
Title: Vedolizumab Study With Inflammatory Bowel Disease Patients in Germany Documentation of Vedolizumab Induction and Maintenance Therapy in Conjunction With Long-term Outcome and Predictors of Response
Brief Title: Vedolizumab Study With Inflammatory Bowel Disease Patients in Germany
Acronym: VEDOibdI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ced Service GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1.4
Record Dates: First submitted 2017-11-06; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Inflammatory Bowel Diseases; Treatment
Keywords: Vedolizumab, Crohns disease, Ulcerative colitis, safety
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1st subpopulation: IBD-patients (age at enrollment: 18-80 years) receiving a newly introduced Vedolizumab (VDZ) therapy (n=1.800). A former therapy with other biologics is allowed. More than 30% of these Vedolizumab patients will be biologics-naiv.
  Interventions: Biological: vedolizumab
- 2nd subpopulation: IBD-patients (age at enrollment: 18-80 years) receiving a newly introduced anti-TNF-alpha therapy other than VDZ (n=350) in biologics-naiv patients.
- 3rd subpopulation: IBD patients (age at enrollment: 18-80 years) with an early disease (n=350), who were first diagnosed <2 years before the start of documentation in the Investigator initiated non-interventional study (NIS) but have not yet received and are not planned to receive biologics in the near future.

INTERVENTIONS:
Biological: vedolizumab — duration of disease and kind of therapy
  Groups: 1st subpopulation

SUMMARY:
This study on biologics (Vedolizumab/anti-TNF) in the treatment of inflammatory bowel disease (IBD) patients in Germany extends the prospective documentation of efficacy in induction and maintenance therapy of anti-TNF to the use of Vedolizumab with a particular interest in the construction of a multifactorial model to predict long-term responses and favorable disease outcome or to predict severe side effects caused by therapy with biologics. Little data are available on the efficacy and safety of biologics in Germany in a real world situation. While the increasing use of anti-TNF-alpha antibodies in IBD-patients the new therapy with Vedolizumab opens up new opportunities in IBD-therapy, it may also pose new options and problems in terms of efficacy and predictors of response and potential side effects.

DETAILED DESCRIPTION:
The IBD-patients will be prospectively documented in the BIOibd-Registry. The diagnosis is made in accordance with current DGVS/ECCO UC/CD guidelines. There are the following inclusion and exclusion criteria:

Inclusion Criteria:

* IBD-patients (UC/CD) aged 18-80 years at enrollment
* Written informed consent is given Exclusion Criteria:Lack of adequate documentation possibilities
* Malignant disease in history
* Planned surgical intervention

There are three subpopulations:

1. IBD-patients (age at enrollment: 18-80 years) receiving a newly introduced Vedolizumab (VDZ) therapy (n=1.800). A former therapy with other biologics is allowed. More than 30% of these Vedolizumab patients will be biologics-naiv.
2. IBD-patients (age at enrollment: 18-80 years) receiving a newly introduced anti-TNF-alpha therapy other than VDZ (n=350) in biologics-naiv patients.
3. IBD patients (age at enrollment: 18-80 years) with an early disease (n=350), who were first diagnosed < 2 years before the start of documentation in the Investigator initiated non-interventional study (NIS) but have not yet received and are not planned to receive biologics in the near future.

Patients with IBD on Vedolizumab/anti-TNF will be documented in a prospective online documentation form at the participating study sites. In parallel, these sites will also document consecutively early disease IBD patients who were diagnosed less than 2 years previously. These patients will be used as a control group.The data will be documented in an online documentation form. After initial documentation at enrollment and during induction (0, 2, 6 and 14 weeks), follow-up documentation using an abbreviated online follow-up form will be requested every 6 months during the longitudinal investigation. Any drug side effects are also captured online on a side effects form.

ELIGIBILITY:
Inclusion Criteria:

* IBD-patients (UC/CD) aged 18-80 years at enrollment
* Written informed consent is given

Exclusion Criteria:

* Lack of adequate documentation possibilities
* Malignant disease in history
* Planned surgical intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are three subpopulations:
  1. IBD-patients (age at enrollment: 18-80 years) receiving a newly introduced Vedolizumab (VDZ) therapy (n=1.800). A former therapy with other biologics is allowed. More than 30% of these Vedolizumab patients will be biologics-naiv.
  2. IBD-patients (age at enrollment: 18-80 years) receiving a newly introduced anti-TNF-alpha therapy other than VDZ (n=350) in biologics-naiv patients.
  3. IBD patients (age at enrollment: 18-80 years) with an early disease (n=350), who were first diagnosed <2 years before the start of documentation in the Investigator initiated non-interventional study (NIS) but have not yet received and are not planned to receive biologics in the near future.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
safety index (Chronic steroid-use ≥ 20 mg for ≥ 6 months, New secreting fistula, Op caused by stenosis, Mortality (all), Hospitalization > 14 days, Long-term-illness (with > 30 days off work), Early retirement) | through study completion, an average of 1 year
  Success - no; Failure - yes

SECONDARY OUTCOMES:
Comparison of the disease course in IBD-patients on Vedolizumab/anti-TNF therapy with IBD-patients with an early-stage disease | during the first 14 weeks after individual participation
  percent responders/remitters at week 2, 6 and 14, time to response, time to remission etc.
Development of a multifactorial model to predict a favorable course of disease | through study completion, an average of 1 year
  Controlling the systematic analysis (e.g. Chronic steroid-use ≥ 20 mg for ≥ 6 months, new secreting fistula etc.) to forecast the good treatment of the participants (to avoid the primary outcome and to reach the secondary outcome/remission).
Online documentation of effectiveness in induction and maintenance therapy including the occurrence of serious side effects | through study completion, an average of 1 year
  Online documentation of effectiveness in induction and maintenance therapy including the occurrence of serious side effects (e.g. death, tumor, tuberculosis, serious infection or other side effects requiring hospitalization.
Efficacy (remission and response) of induction therapy (week 14) | through study completion, an average of 1 year
  Efficacy (remission and response) of induction therapy (week 14)
Generation of health economic data in IBD-patients on biologicals | through study completion, an average of 1 year
  Generation of health economic data in IBD-patients on biologicals (number of hospitalizations, kind of disabilties, cost of treatment, quality of life e.g. WPAI-CD or EQ-5D) through CRF.
Generation of follow-up data on IBD-patients with early disease | through study completion, an average of 1 year
  Generation of follow-up data on IBD-patients with early disease (initiation of documentation < 2 years after first diagnosis) through CRF (e.g. actual diagnostic findings or laboratory reports) and IBD-patients on biologics e.g. actual diagnostic findings or laboratory reports) with reference to treatment modalities and psychosocial impairment among patients.
Formation of a large-scaled patient-collective of IBD-patients with an early course of disease | through study completion, an average of 1 year
  Formation of a large-scaled patient-collective of IBD-patients (350 patients) with an early course of disease (disease course < 2 years) by combining different registries running on the BIOibd platform (6000 patients) of the IBD Competence Net in Germany for the comparison of special subgroups, e.g. IBD-patients on biologics.
Efficacy (remission and response) of maintenance therapy (month 6 and 12) | through study completion, an average of 1 year
  maintenance therapy (month 6 and 12)
Efficacy (remission and response) of effectiveness in different subpopulations | through study completion, an average of 1 year
  effectiveness in different subpopulations, e.g. based on prior biological therapy (remission: HBI ≤ 4 in CD and partial Mayo Score ≤ 1 plus a bleeding subscore of 0 in UC)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Bokemeyer, PD Dr. med., Principal Investigator — Gastroenterologische Gemeinschaftspraxis Minden, Uferstr. 3, 32423 Minden
Locations (1):
- Gastroenterologische Gemeinschaftspraxis Minden, Minden, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No